CLINICAL TRIAL: NCT03831906
Title: Impact of Systematic Early Tuberculosis Detection Using Xpert MTB/RIF Ultra in Children With Severe Pneumonia in High Tuberculosis Burden Countries
Brief Title: Impact of Systematic Early Tuberculosis Detection Using Xpert MTB/RIF Ultra in Children With Severe Pneumonia in High Tuberculosis Burden Countries (TB-Speed Pneumonia)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: C18-26
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis; Severe Pneumonia; Covid19
MeSH Terms: conditions — Tuberculosis; Pneumonia; COVID-19

STUDY DESIGN:
Intervention Model Description: The TB-Speed Pneumonia study is a stepped wedge cluster-randomised trial. Clusters, i.e.hospitals, will successively switch from control to intervention in an order randomly assigned, until all clusters are eventually exposed to the intervention.
  The TB-Speed Pneumonia study will be implemented in 15 hospitals. At the start of the study, all hospital will be implementing the WHO SOC for severe pneumonia (control arm). One hospital will then switch to the TB-Speed strategy (intervention arm) every 5 weeks.
  Randomisation will be stratified on the country estimated TB incidence rate (see Table 3): <300/100,000 patients-years (Cameroon, Cote d'Ivoire and Uganda) vs. ≥300/100,000 patients-years (Cambodia, Mozambique and Zambia).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): All children admitted in the hospital and presenting with WHO-defined severe pneumonia will be immediately managed as part of routine care per the WHO Standard of Care (SOC), including broad spectrum antibiotics, oxygen therapy if required, additional supportive care and specific therapies for comorbidities such as HIV infection.
  For research purposes, children will benefit from HIV testing, malaria testing, and complete blood count (CBC) if not systematically performed as routine care in the country/hospital, as well as from a digitalized chest X-ray (CXR). Additionally, samples will be collected for future biomarkers studies (biobank).
- Interventional (Experimental): Children will benefit from the WHO SOC and additional strategies for research purposes (HIV and malaria testing, CBC, CXR, and biobank) as described in the control arm, plus the study intervention.
  Interventions: Diagnostic Test: Xpert MTB/RIF Ultra (Ultra)

INTERVENTIONS:
Diagnostic Test: Xpert MTB/RIF Ultra (Ultra) — The intervention will consist of the WHO standard of care for children with severe pneumonia plus the study intervention consisting in rapid detection of TB on the day of hospital admission using the Ultra assay performed on 1 NPA and 1 stool sample.
  The sample flow will be organised to reduce time-to-results to 3 hours. Ultra will be performed at the hospital laboratory using a standard GeneXpert device, or implemented directly inward using a one-module, battery-operated GeneXpert device (G1 Edge).
  Drugs will be available at the inpatient level to enable immediate initiation of TB treatment, as soon as a positive Ultra result is available.
  Arms: Interventional

SUMMARY:
Despite progress in reducing tuberculosis (TB) incidence and mortality in the past 20 years, TB is a top ten cause of death in children under 5 years worldwide. However, childhood TB remains massively underreported and undiagnosed, mostly because of the challenges in confirming its diagnosis due to the paucibacillary nature of the disease and the difficulty in obtaining expectorated sputum in children.

Pneumonia is the leading cause of death in children under the age of 5 years worldwide. There is growing evidence that, in high TB burden settings, TB is common in children with pneumonia, with up to 23% of those admitted to hospital with an initial diagnosis of pneumonia later being diagnosed as TB. However, the current World Health Organization (WHO) standard of care (SOC) for young children with pneumonia considers a diagnosis of TB only if the child has a history of prolonged symptoms or fails to respond to antibiotic treatments. Hence, TB is often under-diagnosed or diagnosed late in children presenting with pneumonia.

In this context, the investigators are proposing to assess the impact on mortality of adding the systematic early detection of TB using Xpert MTB/RIF Ultra, performed on NPAs and stool samples, to the WHO SOC for children with severe pneumonia, followed by immediate initiation of anti-TB treatment in children testing positive on any of the samples.

TB-Speed Pneumonia is a multicentric, stepped wedge diagnostic trial conducted in six countries with high TB incidence: Cote d'Ivoire, Cameroon, Uganda, Mozambique, Zambia and Cambodia.

The sub-study on Covid-19 will assess the prevalence and impact of the Covid-19 in young children hospitalized with severe pneumonia. The sub-study findings are expected to guide policy makers and clinicians on potential specific screening and management measures for these vulnerable groups of children. They are also key to analysing TB-Speed Pneumonia results on mortality in a context of the Covid-19 outbreak and to take into consideration SARS-CoV-2 infection status in the main study analysis.

DETAILED DESCRIPTION:
Pneumonia is the leading cause of death in children under the age of 5 years worldwide.

There is growing evidence that, in high TB burden settings, TB is common in children with pneumonia, with up to 23% of those admitted to hospital with an initial diagnosis of pneumonia later being diagnosed as TB]. This is particularly true in the African and Asian WHO regions, which accounted for 30% and 35% of all paediatric TB cases in 2016 respectively.

In these regions, the case fatality rate for childhood pneumonia associated with TB is high, ranging from 4% to 21% [8], with younger age, malnutrition and HIV infection increasing the risk of death.

The current standard of care (SOC) for young children with pneumonia considers a diagnosis of TB only if the child has a history of prolonged symptoms or fails to respond to antibiotic treatments. Hence, TB is often under-diagnosed or diagnosed late in children presenting with pneumonia. Although TB is a chronic disease in adults, recent data show that the duration of respiratory symptoms before admission can be acute in children with severe pneumonia associated with TB [8]. Hence, Identifying TB cases early and shortening the diagnostic delay to initiate appropriate TB treatment in children with clinical presentation of severe acute pneumonia is likely to reduce mortality.

An improved molecular diagnostic tool for paediatric TB:

Xpert MTB/RIF (Cepheid, USA) is an automated nucleic acid amplification test (NAAT) that simultaneously detects Mycobacterium tuberculosis (MTB) and genes associated with resistance to rifampicin. The assay was a major breakthrough in bringing molecular tests for the diagnosis of TB closer to the community, with performances close to mycobacterial culture. WHO therefore recommended Xpert MTB/RIF as the first test to be used for the diagnosis of TB among populations who may have drug-resistant and/or HIV-associated TB.

In 2013, WHO updated its policy to include Xpert MTB/RIF as the initial test for the diagnosis of TB in children, based on a systematic review and meta-analysis showing a pooled sensitivity of 66% (CI 95% 51-81) and a specificity of 98% (CI 95% 96-99) of Xpert MTB/RIF performed on gastric lavages when compared with culture. WHO recommendations, detailed in the 2014 guidance on paediatric TB, stated that Xpert MTB/RIF may be used instead of smear microscopy in all children and should be used in children with HIV infection or presumptive multidrug-resistant TB.

Although data on the performance of Xpert MTB/RIF in children with pneumonia is limited, in Bangladesh, sensitivity on gastric aspirates or sputum samples compared to culture in this group was equivalent to that reported in other studies.

The next-generation of Xpert MTB/RIF assay, Xpert MTB/RIF Ultra (Ultra), has a limit of detection of 16 colony forming units (CFU)/mL (compared to the current version which detects 130 CFU/mL), representing an approximately 8-fold improvement. This lower threshold is similar to the detection level of culture and would facilitate the rapid diagnosis of paucibacillary TB disease as seen in children. Retrospective analyses on frozen respiratory samples in children have shown a sensitivity of 71% for Ultra versus 47% for Xpert MTB/RIF. A recently published study reveals, however, a lower specificity of U ltra in adults, particularly in those with a previous history of TB, potentially resulting in false diagnoses and overtreatment of TB. Though further prospective studies are needed, the risk of false-positive results could be less significant in children as only a small proportion of children have previously had TB. The estimated clinical impact of Ultra is therefore likely to vary depending on the settings, with a recent modelling exercise finding a larger mortality benefit in patient populations with high TB prevalence, high HIV prevalence, and high case fatality ratios for untreated TB.

The current WHO recommendations for the use of Xpert MTB/RIF also apply to the use of Ultra as the initial diagnostic test for all adults and children with signs and symptoms of TB. An update of the current guidelines for the use of Ultra is planned for 2018.

Alternative specimen collection methods adapted to children:

Young children are frequently unable to expectorate sputum and there is no clear evidence and guidance on which specimen or combination of specimens should be used in order to maximize the probability of bacteriological confirmation of TB in children. At the programmatic level, implementation of gastric aspirates and induced sputum can be challenging].

Our research group and other groups in Africa and Asia have shown that alternative specimen collection methods such as nasopharyngeal aspirates (NPA) and stool samples are easier to be implemented in resource-limited settings and are better tolerated in young and sick children. These methods do not require a child to fast (as for gastric aspirates) and are more suitable than induced sputum in children with severe respiratory deficit. In children with presumptive TB, Xpert MTB/RIF has a sensitivity on NPAs close to the one achieved with induced sputum [28], [35]. Recent studies have shown similar sensitivity of Xpert MTB/RIF on the combination of one stool and one NPA as compared to two induced sputum or two gastric aspirates. Stool testing by Xpert MTB/RIF shows results close to respiratory samples in terms of sensitivity but requires a simplified specimen processing methodology for further field use. The flotation method, based on Sheather's sucrose solution used in the PAANTHER study, showed promising results but relies on centrifugation and other labour-intensive processes. Stool processing will be further optimized in Output 4 of the TB-Speed project to enable implementation at a lower healthcare level.

Most studies on childhood TB diagnostics are early proof-of-concepts or studies that evaluate diagnostic accuracy, collecting and testing multiples samples using existing microbiological tests. Implementation studies, with patient health outcomes as the primary endpoint of interest, are seldom implemented despite the need for such studies to inform policies. The WHO recommendation to use Xpert MTB/RIF in children was based on diagnostic accuracy, but evidence of its impact on TB outcome has not been evaluated. As in adults, its use in children may have a limited impact on outcome in children with a strong suspicion of TB, due to the common use of empirical treatment in these populations [48]-[51]. However, this is likely to be different in children with severe pneumonia presenting with acute symptoms, for which TB is usually suspected only after empiric antibiotic treatment has been shown to be ineffective.

The TB-Speed approach to early detection of TB in children with severe pneumonia:

In line with the strategies advocated by the National Tuberculosis Programmes (NTPs) in participating countries, the TB-Speed project aims not only to contribute to the reduction of TB-associated mortality, but also to initiate an innovative approach for the early detection and treatment of TB in young children with severe pneumonia to enable access to high-quality healthcare in this highly vulnerable group.

Our hypothesis is that in high TB burden countries, testing young children with severe pneumonia for TB and starting those who test positive on anti-TB treatment on the day of presentation, could reduce all-cause mortality through reduction of mortality attributed to TB. In this context, the investigators are proposing a research study to assess the impact on mortality of adding the systematic early detection of TB using Ultra performed on NPAs and stool samples to the WHO SOC for children with severe pneumonia, followed by immediate initiation of anti-TB treatment in children testing positive on any of the samples. If successful, this intervention could be systematically implemented at district hospital level where children with severe pneumonia are referred. Furthermore, the investigators hypothesize that the intervention will raise TB awareness among clinicians and may lead to more empirical TB treatment initiated as compared to the control. This further justifies the stepped-wedge design chosen for this study.

From a health economics perspective, the investigators hypothesize that benefits in terms of survival and Disability Adjusted Life Years (DALYs) will outweigh extra costs incurred by systematic Ultra testing in children with severe pneumonia.

Mortality in children aged 2 to 59 months hospitalized with severe pneumonia and mortality attributable to TB:

There were an estimated 120 million pneumonia episodes in children younger than 5 years in 2011, including 14 million severe episodes. 1.3 million pneumonia episodes led to death. In 2014, WHO revised definitions for pneumonia and severe pneumonia, considering 'chest-indrawing pneumonia' as non-severe and downgrading 'pneumonia with severity signs' from very severe to severe. Ambulatory care and oral antibiotics are now recommended for 'chest-indrawing pneumonia' and now only severe pneumonia justifies referral from primary health centres to district hospitals for intra-venous (IV) antibiotics and oxygen therapy if needed.

Participating countries and added value of the multi-country aspect:

The impact of this innovative approach may vary with TB incidence as well as some geographical and seasonal variability that can affect the prevalence and aetiology of pneumonia in young children. To provide a better basis for the generalizability of results, the project will take place in six countries with different epidemiological and environmental backgrounds, in Sub-Saharan Africa (Cameroon, Cote d'Ivoire, Mozambique, Uganda, and Zambia) and South East Asia (Cambodia). Cambodia, Zambia and Mozambique are among the 30 high TB burden countries according to WHO classification.

The sub-study on Covid-19 will assess the prevalence and impact of the Covid-19 in young children hospitalized with severe pneumonia. The sub-study findings are expected to guide policy makers and clinicians on potential specific screening and management measures for these vulnerable groups of children. They are also key to analysing TB-Speed Pneumonia results on mortality in a context of the Covid-19 outbreak and to take into consideration SARS-CoV-2 infection status in the main study analysis. The sub-study will be implemented in all participating countries except Cambodia.

At the time of enrolment in the TB-Speed Pneumonia main study, patients will be also offered to participate to the Covid ancillary study. Children will be tested for SARS-Cov-2 on the day of enrolment. The duration of enrolment in the sub-study will be of 6 months in total. Duration of follow-up for a particular participant will be 12 weeks, as in the main Pneumonia study.

ELIGIBILITY:
Inclusion criteria:

1. Children aged 2 to 59 months
2. Newly hospitalized for severe pneumonia defined using WHO criteria as cough or difficulty in breathing with:

   1. Peripheral oxygen saturation < 90% or central cyanosis, or
   2. Severe respiratory distress (e.g. grunting, nasal flaring, very severe chest indrawing), or
   3. Signs of pneumonia, defined as cough or difficulty in breathing with fast breathing (tachypnea) and/or chest indrawing, with any of the following danger signs:

      * Inability to breastfeed or drink,
      * Persistent vomiting
      * Lethargy or reduced level of consciousness
      * Convulsions,
      * Stridor in calm child
      * Severe malnutrition
3. Informed consent signed by parent/guardian

Exclusion criteria:

- Ongoing TB treatment or history of intake of anti-TB drugs in the last 6 months

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2570 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality 12 weeks after inclusion | 12 weeks

SECONDARY OUTCOMES:
Number of children diagnosed with TB at 12 weeks | 12 weeks
  • Number of children diagnosed with TB at 12 weeks:
  * based on Ultra results
  * based on the clinician's judgement
• Proportion of children with TB treatment initiated at any time during follow-up | 12 weeks
• Time to TB treatment initiation | 12 weeks
• Duration of TB treatment at end of trial | 12 weeks
  • Duration of TB treatment at end of trial, i.e. week 12 or early termination
• Number of inpatient deaths | 12 weeks
• Duration of initial hospitalization | 12 weeks
• Number of readmissions following discharge | 12 weeks
• Weight gain at 12 weeks | 12 weeks
  • Weight gain at 12 weeks, as compared to body weight at inclusion
• Proportion of NPA and stool samples with positive TB detection using Ultra• | 12 weeks
  In the intervention arm only.
• Proportion of Ultra-confirmed and clinically-diagnosed TB cases | 12 weeks
  In the intervention arm only.
• Feasibility of NPA and stool samples collection (1) | 12 weeks
  In the intervention arm only. Proportion of children with samples collected as per protocol
• Feasibility of NPA and stool samples collection (2) | 12 weeks
  In the intervention arm only. Turnaround time between NPA or stool sample collection and result of Ultra
• Safety of NPA collection | 12 weeks
  In the intervention arm only. Adverse events collected by study nurses during NPA collection such as vomiting, nose bleeding, low oxygen saturation
• Tolerability of NPA specimen collection procedures assessed by the child | Hospital admission
  In the intervention arm only. Discomfort/pain/distress experienced by the child assessed by the child him/herself (Wong-Baker face scale)
• Tolerability of NPA specimen collection procedures assessed by the parents | Hospital admission
  In the intervention arm only. Discomfort/pain/distress experienced by the child assessed by the parents (visual analog scale)
• Tolerability of NPA specimen collection procedures assessed by the nurses | Hospital admission
  In the intervention arm only. Discomfort/pain/distress experienced by the child assessed by the nurses (FLACC behavioural scale)
• Acceptability of NPA and stool specimen collection procedures | Hospital admission
  In the intervention arm only.
  • Acceptability of NPA and stool specimen collection procedures assessed by parents and nurses (semi-structured interviews and auto-questionnaires).
To assess the prevalence of Covid-19 (confirmed and probable cases) in children below 5 years admitted with WHO-defined severe pneumonia | 12 weeks
Number of inpatients death in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 12 weeks
Duration of initial hospitalization in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 12 weeks
Number of readmissions following discharge in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 12 weeks
Weight gain in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 12 weeks
Inability to breastfeed or drink in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Inability to breastfeed or drink in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Inability to breastfeed or drink in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Lethargy or reduced level of consciousness in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Lethargy or reduced level of consciousness in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Lethargy or reduced level of consciousness in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Convulsions in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Convulsions in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Convulsions in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Stridor in calm child in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Stridor in calm child in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Stridor in calm child in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Oxygen saturation < 90% in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Oxygen saturation < 90% in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Oxygen saturation < 90% in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Central cyanosis in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Central cyanosis in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Central cyanosis in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Grunting in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Grunting in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Grunting in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Nasal flaring in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Nasal flaring in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Nasal flaring in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
Chest in-drawing in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | Hospital admission
Chest in-drawing in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | 3 day after hospitalisation
Chest in-drawing in children with severe pneumonia (infected with SARS-CoV-2 versus to uninfected children) | At hospital discharge, estimated average = 7 days
To describe the laboratory characteristics (CRP) of Covid-19 cases | 12 weeks
To describe the laboratory characteristics (full blood count) of Covid-19 cases | 12 weeks
Description by type and frequency of the signs of viral pneumonia on CXR with interstitial changes of Covid-19 cases | 12 weeks
To assess the yield of stool as compared to nasal swab for the detection of the SARS-CoV-2 by real time reverse transcription-polymerase chain reaction (RT-PCR) | 12 weeks
Number of children having a PCR positive for respiratory syncytial virus | 12 weeks
  PCR detection of respiratory syncytial virus
To assess seroprevalence and seroconversion (immunoglobulin M and immunoglobulin G to SARS-CoV-2) at Day 0 and Month 3 | 12 weeks

OTHER OUTCOMES:
Comparison of the cost-effectiveness of the two strategies | 12 weeks
  Incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, MD, PhD, Principal Investigator — University of Bordeaux, France; Maryline Bonnet, MD, PhD, Principal Investigator — Institut de Recherche pour le Développemnt (IRD) Montpellier, France; Eric Wobudeya, MD, PhD, Principal Investigator — MU-JHU Care Ltd, Kampala, Uganda
Locations (16):
- Cambodia (3):
  - Kampong Cham Provincial Referral Hospital, Kampong Cham
  - National Pediatric Hospital, Phnom Penh
  - Takeo Provincial Referral Hospital, Takeo
- Cameroon (2):
  - Biyem Assi District Hospital, Yaoundé
  - Chantal Biya Foundation, Yaoundé
- Côte d’Ivoire (4):
  - Angré University Teaching Hospital, Abidjan
  - Cocody University Teaching Hospital, Abidjan
  - Treichville University Teaching Hospital, Abidjan
  - Yopougon University Teaching Hospital, Abidjan
- Mozambique (2):
  - José Macamo General Hospital, Maputo
  - Maputo Central Hospital, Maputo
- Uganda (3):
  - Jinja Regional Reference Hospital, Jinja
  - Mulago National Referral Hospital, Kampala
  - Holy Innocents Children's Hospital, Mbarara
- Zambia (2):
  - Lusaka University Teaching Hospital, Lusaka
  - Arthur Davidson Children Hospital, Ndola

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Vessiere A, Font H, Gabillard D, Adonis-Koffi L, Borand L, Chabala C, Khosa C, Mavale S, Moh R, Mulenga V, Mwanga-Amumpere J, Taguebue JV, Eang MT, Delacourt C, Seddon JA, Lounnas M, Godreuil S, Wobudeya E, Bonnet M, Marcy O. Impact of systematic early tuberculosis detection using Xpert MTB/RIF Ultra in children with severe pneumonia in high tuberculosis burden countries (TB-Speed pneumonia): a stepped wedge cluster randomized trial. BMC Pediatr. 2021 Mar 20;21(1):136. doi: 10.1186/s12887-021-02576-5. PMID 33743621
- [Derived] Marcy O, Wobudeya E, Font H, Vessiere A, Chabala C, Khosa C, Taguebue JV, Moh R, Mwanga-Amumpaire J, Lounnas M, Mulenga V, Mavale S, Chilundo J, Rego D, Nduna B, Shankalala P, Chirwa U, De Lauzanne A, Dim B, Tiogouo Ngouana E, Folquet Amorrissani M, Cisse L, Amon Tanoh Dick F, Komena EA, Kwedi Nolna S, Businge G, Natukunda N, Cumbe S, Mbekeka P, Kim A, Kheang C, Pol S, Maleche-Obimbo E, Seddon JA, Mao TE, Graham SM, Delacourt C, Borand L, Bonnet M; TB-Speed Pneumonia Study Group. Effect of systematic tuberculosis detection on mortality in young children with severe pneumonia in countries with high incidence of tuberculosis: a stepped-wedge cluster-randomised trial. Lancet Infect Dis. 2023 Mar;23(3):341-351. doi: 10.1016/S1473-3099(22)00668-5. Epub 2022 Nov 14. PMID 36395782
- [Derived] Kay AW, Gonzalez Fernandez L, Takwoingi Y, Eisenhut M, Detjen AK, Steingart KR, Mandalakas AM. Xpert MTB/RIF and Xpert MTB/RIF Ultra assays for active tuberculosis and rifampicin resistance in children. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD013359. doi: 10.1002/14651858.CD013359.pub2. PMID 32853411
- See also: TB-Speed project official website — https://www.tb-speed.com